CLINICAL TRIAL: NCT04212780
Title: Dual Lead Thalamic DBR-DBS Interface for Closed Loop Control of Severe Essential Tremor
Brief Title: Dual Lead Thalamic Deep Brain Recording (DBR)-DBS Interface for Closed Loop Control of Severe Essential Tremor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: IRB201901021; OCR29622 (Other: University of Florida); 1UH3NS109845-01 (NIH); 5UH3NS109845-02 (NIH)
Record Dates: First submitted 2019-12-19; First posted 2019-12-30 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-08

CONDITIONS: Essential Tremor
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment Naive (Active Comparator): Participants receiving Long-term stimulation of the thalamus via dual leads for Essential Tremor
  Interventions: Device: Medtronic Summit Rechargable (RC)+S; Procedure: standard ET DBS; Procedure: ipsilateral VO
- Refractory Participants (Active Comparator): Patients with recurrent, debilitating intention tremor despite ongoing, optimized VIM DBS therapy
  Interventions: Device: Medtronic Summit Rechargable (RC)+S; Procedure: ipsilateral thalamic (VIM+VO) DBS

INTERVENTIONS:
Device: Medtronic Summit Rechargable (RC)+S — Dual channel closed-loop pulse generator with connection to both new DBS leads for deep stimulation of VIM vs VO
Procedure: ipsilateral thalamic (VIM+VO) DBS — Implantation of two new ipsilateral thalamic (VIM+VO) DBS
  Arms: Refractory Participants
Procedure: standard ET DBS — Single Lead VIM
  Arms: Treatment Naive
Procedure: ipsilateral VO — second lead in the ipsilateral VO
  Arms: Treatment Naive

SUMMARY:
This is a feasibility study based on physician-initiated Investigational Device Exemption (IDE) including intraoperative experiments and chronic testing of implanted dual thalamic DBS lead systems. This study will inform protocols for optimal use of implanted next-gen DBS systems for primarily tremor control in refractory essential tremor.If the approach appears to be successful, the pilot data generated will be used to base a future pivotal trial for FDA approval for enhanced tremor control and adaptive DBS (aDBS) functionality of DBS systems.

DETAILED DESCRIPTION:
Ventralis intermedius nucleus of the thalamus (VIM) Deep Brain Stimulation (DBS) has emerged as a highly effective treatment for essential tremor, which is an incurable, degenerative brain disorder that results in progressively debilitating tremor, afflicting an estimated 7 million people in the US (2.2% of the population). Clinical observation shows, however, that disease progression results in eventual recurrence of debilitating tremor in 10 to 20% of VIM DBS patients. DBS revision surgery, with replacement of sub-optimally positioned VIM DBS leads and addition of an ipsilateral ventralis oralis (VO) DBS lead, has emerged as an effective rescue strategy for many such patients with delayed failure of VIM DBS therapy.

Since essential tremors are typically not continuous, tremor suppressing DBS therapy need not necessarily be delivered continuously and could theoretically be effective if delivered only when movement intent or tremor is present.

Our central hypothesis is that a VIM+VO DBS system capable of detecting the neurophysiologic markers of essential tremor (ET) associated with goal directed movements, and providing responsive dual lead thalamic stimulation in a targeted and personalized manner, would provide improved suppression of severe tremor, reduce adverse effects associated with continuous stimulation, and prolong the battery life of the implantable neurostimulator (INS), decreasing the frequency of surgical procedures necessary to replace devices with depleted batteries.

ELIGIBILITY:
Inclusion Criteria:

* Patient gives an informed consent.
* Patient is over 21 years of age.
* Patient is diagnosed with a postural-intention (essential) tremor for at least 3 years, meets diagnostic criteria for ET, has been evaluated and examined by a movement disorders fellowship trained neurologist, and is being treated with traditional VIM DBS therapy.
* Patient has no evidence of non-ET central nervous system disease or injury and has had a significantly disabling, upper extremity tremor despite ongoing VIM DBS therapy for at least three (3) months prior to DBS revision surgery.
* Patient has a postural or kinetic tremor severity score of at least 2 out of 4 in the extremity intended for treatment on the Fahn-Tolosa-Marin Clinical Rating Scale for Tremor (TRS) despite ongoing VIM DBS therapy.
* Patient has a TRS score of 2 or above in any one of the items 16-23 from the Disability subsection of the TRS: speaking, feeding other than liquids, bringing liquids to mouth, hygiene, dressing, writing, working and social activities despite ongoing VIM DBS therapy.
* Patient's tremor is refractory to adequate trials of at least two medications, one of which should be either propranolol or primidone. Proof of this is not required for patients with a current device that is being removed and replaced with a new device. An adequate medication trial is defined as a therapeutic dose of each medication or the development of side effects as the medication dose is titrated.
* Patient is available for appropriate follow-up times for the length of the study.

Exclusion Criteria:

* Any previous neurosurgical intervention other than VIM DBS, including ablative brain lesions for tremor suppression.
* Medication related movement disorders.
* Any suspicion of Parkinson's disease, including presence of Parkinsonian features such as bradykinesia, rigidity, or postural instability.
* Any behaviors consistent with alcohol or substance abuse as defined by the criteria outlined in Diagnostic and Statistical Manual of Mental Disorders (DSM-V).
* Severe medical co-morbidity including cardiovascular disorder, lung disorder, kidney disease, continuous neurological disease, hematological disease, or frailty that impact tolerability of the surgery as judged by the screening physicians.
* Abnormal brain MRI including hydrocephalus, stroke, structural lesions, demyelinating lesions, or infectious lesions. Also excluded will be subjects with severe brain atrophy.
* Any uncontrolled symptoms or signs of increased intracranial pressure (e.g., headache, nausea, vomiting, lethargy, papilledema).
* A history of seizures within the past year.
* A dementia rating scale score (DRS) <130 signifying significant cognitive dysfunction and a potential for inability to cooperate with tasks involved in the study.
* Any attempt or intent of suicide during the previous six months.
* Presence or history of psychosis.
* Any person known to have abnormal coagulation or any medications which interfere with coagulation
* Significant untreated or unstable mood disorders including depression. This will be determined by the Neuropsychological team during FastTrack and by the Neurologist
* In addition, patients who are pregnant or plan to become pregnant will be excluded from this study.

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-12-24 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy Assessment - Tremor | Up to 24 months
  Tremor rating scale This 5-point scale rates tremor severity based on tremor amplitude, from 0 (no tremor) to 4 (severe tremor) in each part of the body, and includes assessments of specific abilities and functional disability.

CONTACTS AND LOCATIONS:
Overall Officials: Karim Oweiss, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No